CLINICAL TRIAL: NCT02030015
Title: Synergistic Enteral Regimen for Treatment of the Gangliosidoses (Syner-G)
Brief Title: Synergistic Enteral Regimen for Treatment of the Gangliosidoses
Acronym: Syner-G
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Efficacy
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Lysosomal Disease Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Syner_G_Regimen; U54NS065768 (NIH); 1311M46101 (Other: Univ. of Minnesota IRB Identifier Number)
Record Dates: First submitted 2013-12-17; First posted 2014-01-08 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: GM1 Gangliosidoses; GM2 Gangliosidoses; Tay-Sachs Disease; Sandhoff Disease
Keywords: infantile Tay-Sachs disease; juvenile Tay-Sachs disease; infantile GM1 gangliosidosis; juvenile GM1 gangliosidosis; infantile GM2 gangliosidosis; juvenile GM2 gangliosidosis; Sandhoff disease; gangliosidoses; miglustat; ketogenic diet; SYNER-G regimen; Syner-G; Zavesca; Tay-Sachs disease; Tay Sachs disease
MeSH Terms: conditions — Gangliosidoses, GM2; Tay-Sachs Disease; Sandhoff Disease; Tay-Sachs Disease, Juvenile; Gangliosidosis, GM1; Gangliosidoses | interventions — miglustat; Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Syner-G Therapy Regimen (Experimental): The Syner-G therapy regimen includes switching the research subject to a full-time ketogenic diet, and daily treatment with orally-administered miglustat, for the duration of the 60-month study.
  Interventions: Drug: miglustat; Other: Ketogenic Diet

INTERVENTIONS:
Drug: miglustat — The Syner-G therapy regimen includes treating with orally-administered miglustat for the duration of the 60-month study.
  Other Names: Zavesca®
Other: Ketogenic Diet — The Syner-G therapy regimen includes switching the research subject to a full-time ketogenic diet for the 60-month duration of this study.

SUMMARY:
The investigators hypothesize that a combination therapy using miglustat and the ketogenic diet for infantile and juvenile patients with gangliosidoses will create a synergy that 1) improves overall survival for patients with infantile or juvenile gangliosidoses, and 2) improves neurodevelopmental clinical outcomes of therapy, compared to data reported in previous natural history studies. The ketogenic diet is indicated for management of seizures in patients with seizure disorders. In this study, the ketogenic diet will be used to minimize or prevent gastrointestinal side-effects of miglustat. A Sandhoff disease mouse study has shown that the ketogenic diet may also improve central nervous system response to miglustat therapy (see Denny in "Citations" list below). Patients with infantile and juvenile gangliosidoses commonly suffer from seizure disorders, and use of the ketogenic diet in these patients may therefore also improve seizure management.

DETAILED DESCRIPTION:
The infantile and juvenile forms of GM1 and GM2 gangliosidoses are neurodegenerative conditions that are lethal during childhood. There are no known effective therapies available for treatment of infantile and juvenile gangliosidoses. Studies of monotherapy with miglustat for treatment of these conditions have demonstrated safety, but have not demonstrated notable clinical improvement. To date, combination therapy for the infantile and juvenile gangliosidoses has not been explored. This study will evaluate a multi-targeted combination therapy for treatment of the gangliosidoses, using FDA approved therapies that have demonstrated safety in children. It is the aim of this study to learn if combination therapy using the "Syner-G" regimen (that is, synergistic enteral regimen for treatment of the gangliosidoses) will show improvement in overall survival and clinical benefits in neurodevelopmental abilities in children with gangliosidosis diseases.

This study is planned as a 5-year longitudinal treatment study. Subjects will be started on the treatment regimen when they are enrolled in the study. Data will be collected during yearly evaluations and at completion of study. Investigators may choose to stop therapy at any time, as clinically indicated for individual patients.

The Ketogenic Diet is a special diet that contains higher amounts of fat and lower amounts of carbohydrate compared to an average diet. The purpose of this is to help reduce food-miglustat interactions. The ketogenic diet may also help in management of seizures in these patients. (The ketogenic diet has been used as an anti-seizure treatment in a variety of medical conditions for many decades.) A study in Sandhoff disease mice has shown that the ketogenic diet may also help miglustat be more effective in the central nervous system (see Denny in "Citations" list below).

Miglustat will be used to reduce the amount of ganglioside accumulation in the child's cells. Miglustat is not FDA approved for treatment of the gangliosidoses. It is FDA approved for a different inherited metabolic disease called Gaucher disease type I.

This study has been issued Investigational New Drug (IND) # 127636 by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a documented infantile or juvenile gangliosidosis disease.
2. Age: 17 years or less at time of enrollment
3. Subjects and their caregivers must be willing to work with a ketogenic diet team for management of the subject's ketogenic diet.

Exclusion Criteria:

1. A desire to not participate
2. Patients who are older than 17 years will not be enrolled in this study.
3. Children with severe renal impairment will not be enrolled in this study.
4. Post-pubertal females who are pregnant, or who are unwilling to use highly-effective methods to prevent pregnancy, will be excluded from this study.
5. Breast-feeding females will be excluded from this study.
6. Subjects who have an allergy to miglustat or any of the components within the drug product will be excluded from this study.

Max Age: 204 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine R. Jarnes, PharmD, Principal Investigator — University of Minnesota Fairview Hospital
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data is input to the NIH-funded Rare Diseases Clinical Research Network's Data Management & Coordinating Center ("DMCC"). Eventually this data will become part of the database of Genotypes and Phenotypes ("dbGaP"), which is part of the National Center for Biotechnology Information, U.S. National Library of Medicine.

REFERENCES:
- [Background] Bley AE, Giannikopoulos OA, Hayden D, Kubilus K, Tifft CJ, Eichler FS. Natural history of infantile G(M2) gangliosidosis. Pediatrics. 2011 Nov;128(5):e1233-41. doi: 10.1542/peds.2011-0078. Epub 2011 Oct 24. PMID 22025593
- [Background] Nalini A, Christopher R. Cerebral glycolipidoses: clinical characteristics of 41 pediatric patients. J Child Neurol. 2004 Jun;19(6):447-52. doi: 10.1177/088307380401900610. PMID 15446395
- [Background] Maegawa GH, Stockley T, Tropak M, Banwell B, Blaser S, Kok F, Giugliani R, Mahuran D, Clarke JT. The natural history of juvenile or subacute GM2 gangliosidosis: 21 new cases and literature review of 134 previously reported. Pediatrics. 2006 Nov;118(5):e1550-62. doi: 10.1542/peds.2006-0588. Epub 2006 Oct 2. PMID 17015493
- [Background] Maegawa GH, van Giersbergen PL, Yang S, Banwell B, Morgan CP, Dingemanse J, Tifft CJ, Clarke JT. Pharmacokinetics, safety and tolerability of miglustat in the treatment of pediatric patients with GM2 gangliosidosis. Mol Genet Metab. 2009 Aug;97(4):284-91. doi: 10.1016/j.ymgme.2009.04.013. Epub 2009 May 3. PMID 19447653
- [Background] Shapiro BE, Pastores GM, Gianutsos J, Luzy C, Kolodny EH. Miglustat in late-onset Tay-Sachs disease: a 12-month, randomized, controlled clinical study with 24 months of extended treatment. Genet Med. 2009 Jun;11(6):425-33. doi: 10.1097/GIM.0b013e3181a1b5c5. PMID 19346952
- [Background] Belmatoug N, Burlina A, Giraldo P, Hendriksz CJ, Kuter DJ, Mengel E, Pastores GM. Gastrointestinal disturbances and their management in miglustat-treated patients. J Inherit Metab Dis. 2011 Oct;34(5):991-1001. doi: 10.1007/s10545-011-9368-7. Epub 2011 Jul 21. PMID 21779792
- [Background] Kossoff EH, Zupec-Kania BA, Amark PE, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Helen Cross J, Dahlin MG, Donner EJ, Klepper J, Jehle RS, Kim HD, Christiana Liu YM, Nation J, Nordli DR Jr, Pfeifer HH, Rho JM, Stafstrom CE, Thiele EA, Turner Z, Wirrell EC, Wheless JW, Veggiotti P, Vining EP; Charlie Foundation, Practice Committee of the Child Neurology Society; Practice Committee of the Child Neurology Society; International Ketogenic Diet Study Group. Optimal clinical management of children receiving the ketogenic diet: recommendations of the International Ketogenic Diet Study Group. Epilepsia. 2009 Feb;50(2):304-17. doi: 10.1111/j.1528-1167.2008.01765.x. Epub 2008 Sep 23. PMID 18823325
- [Background] Zaroff CM, Neudorfer O, Morrison C, Pastores GM, Rubin H, Kolodny EH. Neuropsychological assessment of patients with late onset GM2 gangliosidosis. Neurology. 2004 Jun 22;62(12):2283-6. doi: 10.1212/01.wnl.0000130498.19019.02. PMID 15210895
- [Background] Bembi B, Marchetti F, Guerci VI, Ciana G, Addobbati R, Grasso D, Barone R, Cariati R, Fernandez-Guillen L, Butters T, Pittis MG. Substrate reduction therapy in the infantile form of Tay-Sachs disease. Neurology. 2006 Jan 24;66(2):278-80. doi: 10.1212/01.wnl.0000194225.78917.de. PMID 16434676
- [Background] Zupec-Kania BA, Spellman E. An overview of the ketogenic diet for pediatric epilepsy. Nutr Clin Pract. 2008 Dec-2009 Jan;23(6):589-96. doi: 10.1177/0884533608326138. PMID 19033218
- [Background] Denny CA, Heinecke KA, Kim YP, Baek RC, Loh KS, Butters TD, Bronson RT, Platt FM, Seyfried TN. Restricted ketogenic diet enhances the therapeutic action of N-butyldeoxynojirimycin towards brain GM2 accumulation in adult Sandhoff disease mice. J Neurochem. 2010 Jun;113(6):1525-35. doi: 10.1111/j.1471-4159.2010.06733.x. Epub 2010 Apr 3. PMID 20374428
- [Background] Utz JR, Crutcher T, Schneider J, Sorgen P, Whitley CB. Biomarkers of central nervous system inflammation in infantile and juvenile gangliosidoses. Mol Genet Metab. 2015 Feb;114(2):274-80. doi: 10.1016/j.ymgme.2014.11.015. Epub 2014 Dec 6. PMID 25557439
- [Background] Karimzadeh P, Naderi S, Modarresi F, Dastsooz H, Nemati H, Farokhashtiani T, Shamsian BS, Inaloo S, Faghihi MA. Case reports of juvenile GM1 gangliosidosisis type II caused by mutation in GLB1 gene. BMC Med Genet. 2017 Jul 17;18(1):73. doi: 10.1186/s12881-017-0417-4. PMID 28716012
- [Background] Deodato F, Procopio E, Rampazzo A, Taurisano R, Donati MA, Dionisi-Vici C, Caciotti A, Morrone A, Scarpa M. The treatment of juvenile/adult GM1-gangliosidosis with Miglustat may reverse disease progression. Metab Brain Dis. 2017 Oct;32(5):1529-1536. doi: 10.1007/s11011-017-0044-y. Epub 2017 Jun 3. PMID 28577204
- [Background] Brackmann F, Kehrer C, Kustermann W, Bohringer J, Krageloh-Mann I, Trollmann R. Rare Variant of GM2 Gangliosidosis through Activator-Protein Deficiency. Neuropediatrics. 2017 Apr;48(2):127-130. doi: 10.1055/s-0037-1598646. Epub 2017 Feb 13. PMID 28192816
- [Background] Regier DS, Proia RL, D'Azzo A, Tifft CJ. The GM1 and GM2 Gangliosidoses: Natural History and Progress toward Therapy. Pediatr Endocrinol Rev. 2016 Jun;13 Suppl 1(Suppl 1):663-73. PMID 27491214
- [Background] Nestrasil I, Ahmed A, Utz JM, Rudser K, Whitley CB, Jarnes-Utz JR. Distinct progression patterns of brain disease in infantile and juvenile gangliosidoses: Volumetric quantitative MRI study. Mol Genet Metab. 2018 Feb;123(2):97-104. doi: 10.1016/j.ymgme.2017.12.432. Epub 2017 Dec 20. PMID 29352662
- [Result] Jarnes Utz JR, Kim S, King K, Ziegler R, Schema L, Redtree ES, Whitley CB. Infantile gangliosidoses: Mapping a timeline of clinical changes. Mol Genet Metab. 2017 Jun;121(2):170-179. doi: 10.1016/j.ymgme.2017.04.011. Epub 2017 Apr 29. PMID 28476546
- See also: Educational information for the layperson about Tay-Sachs disease from the National Organization for Rare Disorders (NORD) — http://rarediseases.org/rare-diseases/tay-sachs-disease/
- See also: Educational information for the layperson about Tay-Sachs disease from the National Human Genome Research Institute at the NIH — https://www.genome.gov/10001220/
- See also: Talking Glossary of Genetic Terms from the National Human Genome Research Institute at the NIH. (Uses Adobe Flash plugin.) This Talking Glossary is also available as an app for mobile devices, from a link on this page. — https://www.genome.gov/glossary/
- See also: Rare Diseases Clinical Research Network, an NIH-funded research network — https://www.rarediseasesnetwork.org/
- See also: The Lysosomal Disease Network's page on the Rare Diseases Clinical Research Network's web site — https://www.rarediseasesnetwork.org/LDN/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Syner-G Therapy Regimen
Started | 16
Completed | 0
Not Completed | 16
Not completed — Withdrawal by Subject | 3
Not completed — Death | 13

BASELINE CHARACTERISTICS:
Arm/Group | Syner-G Therapy Regimen
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: The Duration of Survival of Each Research Subject, Measured in Months and Years
Description: The survival duration of patients with infantile and juvenile forms of gangliosidoses will be assessed, in order to judge the clinical impact of the Syner-G therapy regimen. This will be accomplished by recording the subject's age on the date of enrollment in this study, and the subject's age at the conclusion of this study, or on the date of their death, whichever comes first. The duration of each subject's survival, expressed in months and years, will be compared to available natural history data in order to arrive at an expert assessment of the impact of the Syner-G therapy upon patient longevity.
Time Frame: From date of enrollment until 60 months thereafter, or the date of subject's death from any cause, whichever comes first, assessed up to 60 months
Population: No participants completed the trial. Outcome measure data was not collected due to small sample size.
Arm/Group | Syner-G Therapy Regimen
Number analyzed (Participants) | 0

2. Secondary Outcome: Rate of Change in Neurocognitive Functioning
Description: The Bayley Scales of Infant and Toddler Development and the Vineland Adaptive Behavior Scales will be administered upon enrollment and annually thereafter for five years. Changes in these neurodevelopmental assessments will be evaluated over the duration of follow-up. Ability of the child to have these assessments yearly may be subject to patient's insurance coverage for such assessments.
Time Frame: Upon Enrollment, and thereafter at 12, 24, 36, 48 and 60 months post-enrollment
Population: No participants completed the trial. Outcome measure data was not collected due to small sample size.
Arm/Group | Syner-G Therapy Regimen
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were followed for the length of study participation; up to 60 months or 5 years
Arm/Group | Syner-G Therapy Regimen
All-Cause Mortality (participants affected / at risk) | 13/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT02030015/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02030015/ICF_001.pdf